CLINICAL TRIAL: NCT04922931
Title: Post-COVID 19 Patients Undergoing Surgery: Determination of Residual Lung Abnormalities and Postoperative Adverse Effects
Brief Title: Post-COVID 19 Patients Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)346/2020
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Post-COVID patients; pulmonary sequelae; postoperative complications
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID-19 group: The Post-COVID-19 group or case group includes post-COVID patients (confirmed by PCR) >18 years undergoing scheduled surgery without pulmonary disease prior to SARS-CoV-2 infection that at the time of surgery present negative PCR and absence of clinic due to SARS-CoV-2.
  Interventions: Procedure: scheduled surgery
- Control group: The control group includes patients over the age of 18 who did not have COVID-19 and without moderate-severe pulmonary pathology prior to surgery and in conditions of hemodynamic and respiratory stability at time of surgery.
  Interventions: Procedure: scheduled surgery

INTERVENTIONS:
Procedure: scheduled surgery — Patients undergoing scheduled surgery with lung ultrasound before surgery and determination of lung compliance during general anesthesia

SUMMARY:
More and more patients are undergoing elective surgery after SARS-CoV-2 infection, and little is known about the residual pulmonary changes in these patients after infection and postoperative pulmonary complications. So, we propose an observational study comparing postCOVID-19 patients with normal population (control group) undergoing surgery.

DETAILED DESCRIPTION:
The most common lung complications of severe COVID-19 are pneumonia and hypoxemic respiratory failure/ARDS. Manifestations of lung inflammation or fibrosis were also observed in late stages of COVID-19 causing respiratory sequelae. Fibrous lesions may form during the healing of pulmonary chronic inflammation or proliferative diseases, with gradual replacement of cellular components by scar tissues indicating a poor outcome of COVID-19. Ultrasound allows to stratify the severity of lung damage and combined with the clinic, can help estimate the patient's prognosis and support therapeutic decision-making. On the other hand, pulmonary inflammatory processes and fibrosis are responsible for a decrease in respiratory distensibility or pulmonary compliance. Pulmonary parenchyma distensibility is known as static distensibility or compliance and it´s calculated by mechanical ventilators during general anesthesia.

There are no studies that determine the results of lung ultrasound and pulmonary compliance in preoperative and intraoperative period respectively in postCOVID patients, and the postoperative complications of postCOVID patients are poorly understood.

ELIGIBILITY:
Control group

Inclusion criteria.:

-Patients over the age of 18 who did not have COVID-19 and who are going to undergo scheduled surgery

Exclusion criteria:

* Patients under the age of 18.
* Unstable patients in shock
* Patients in current state of pulmonary hypertension or heart failure
* Patients with moderate-severe pulmonary pathology prior to surgery.
* Patients previously surgery for chest surgery
* Patients in current state of respiratory infection

Post-COVID group Inclusion criteria

-Post-COVID-19 patients (confirmed by PCR) >18 years undergoing scheduled surgery without pulmonary disease prior to SARS-CoV-2 infection, that at the time of surgery present negative PCR and absence of clinic due to SARS-CoV-2 infection.

Exclusion criteria:

* Patients under the age of 18
* Unstable patients in shock
* Patients in current state of pulmonary hypertension or heart failure
* Patients with moderate-severe pulmonary pathology prior to SARS-CoV-2.
* Patients previously surgery for chest surgery
* Patients in current state of respiratory infection

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The written consent forms are obtained from all the subjects who agreed to participate in the study. Patients who suffered Covid-19 prior to surgery without previous moderate-severe pulmonary pathology, that at the time of surgery present negative PCR and absence of clinic due to SARS-CoV-2, are included in the Post-COVID 19 group. The "control group" includes patients over the age of 18 who did not have COVID-19 and without moderate-severe pulmonary pathology prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Determination of residual pulmonary alterations in post-COVID patients | 1 month
  1. Determination of residual pulmonary alterations using preoperative lung ultrasound and obtaining intraoperative compliance in postCOVID-19 patients undergoing surgery.
Correlation between lung ultrasound and pulmonary compliance | 1 month
  Analyze the correlation between the values obtained with pulmonary ultrasound and the pulmonary compliance obtained by mechanical ventilation in patients with general anesthesia.

SECONDARY OUTCOMES:
postoperative complications | 1 month
  Determine postoperative complications one month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Susana González-Suárez, PhD, Principal Investigator — Vall d´Hebron Institut Research (VHIR)
Locations (1):
- Vall d´Hebron Research Institute VHIR, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Suarez S, Barbara Ferreras A, Caicedo Toro M, Aznar de Legarra M. Detection of residual pulmonary alterations with lung ultrasound and effects on postoperative pulmonary complications for patients with asymptomatic SARS-CoV-2 infection undergoing surgeries. BMC Anesthesiol. 2022 Jun 16;22(1):186. doi: 10.1186/s12871-022-01715-4. PMID 35710326